CLINICAL TRIAL: NCT01119872
Title: Randomized Controlled Pilot Study of Positive End-Expiratory Pressure (PEEP) in Acute Respiratory Distress Syndrome(ARDS): Individualized According to the Best Compliance or Fixed According to Fraction of Inspired Oxygen (FiO2) Applied
Brief Title: Pilot Study of Positive-End Expiratory Pressure in Acute Respiratory Distress Syndrome
Acronym: PEEP-HUPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Principe de Asturias (Other)
Responsible Party: María del Consuelo Pintado, Critical Care Unit. Universitary Hospital Príncipe de Asturias
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCI-HUPA-1
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2010-05-10 (Estimated); Status verified 2002-12

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Positive-Pressure Respiration; Respiration, Artificial
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Aspiration | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compliance-guided PEEP group (Other): Positive End-Expiratory Pressure(PEEP) level was set daily, according to the method described by Suter in 1978. Static compliance (Cst) was calculated at different levels of PEEP at a constant tidal ventilation of 6-8 ml/kg of predicted body weight. Cst was determined by dividing tidal volume by the difference between the pressure at the end of inflation hold and the PEEP. The maximum value of Cst in individual patients was considered as the best PEEP.
  Interventions: Other: Positive End-expiratory Pressure (PEEP)
- FiO2-driven-PEEP group (Other): PEEP was set based on the patient fraction of inspired oxygen (FiO2) according to the Positive End-Expiratory Pressure(PEEP) strategy reported in 2000:"Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. The Acute Respiratory Distress Syndrome Network".
  Interventions: Other: Positive End-expiratory Pressure (PEEP)

INTERVENTIONS:
Other: Positive End-expiratory Pressure (PEEP) — All patients were ventilated during 24 hours with low tidal volume (6-8 milliliters/kilogram of predicted body weight), plateau airway pressure limited at 35 centimeters of water, initial ventilator rate of 30 breaths/minute adjusted to maintain a pH goal of 7.30 to 7.45 to a maximum of 35 breaths/minute, fraction of inspired oxygen ensuring arterial oxygen saturation 88-95% or arterial partial pressure of oxygen of 55-80 mmHg.
  Level of Positive End-Expiratory Pressure (PEEP) applied according the 2 arms of treatment.
  Other Names: Compliance-guided PEEP group: Grupo meseta; FiO2-driven-PEEP group: Grupo tabla

SUMMARY:
Randomized controlled pilot trial in 70 patients with Acute Respiratory Distress Syndrome (ARDS) ventilated with low tidal volumes and limitation on airway pressure at 35 centimeters of water (cmH2O), to compare two different methods of selecting the level of Positive End-Expiratory Pressure (PEEP) to be applied: according to fraction of inspired oxygen (FiO2) needed or individualized according to the best compliance. Primary objective was evolution of arterial oxygenation during the 28 days. Secondary objectives were to measure its effects on hemodynamic parameters, 28-day mortality, number of ventilator-free days at day 28, Intensive Care Unit (ICU) and hospital stay, number of multiple-organ dysfunction-free days and a multivariate analysis of 28 day-mortality.

DETAILED DESCRIPTION:
In patients with Acute Respiratory Distress Syndrome the use of Positive End-Expiratory Pressure (PEEP) avoids atelectrauma, improves gas exchange and induces alveolar recruitment.Although it has side effects as inducing alveolar overdistension and circulatory depression.

There are several methods to determine the level of PEEP to be applied. We conducted a study to test the hypothesis that an individualized level of PEEP, set et the best compliance, when compared with a fixed level according to the fraction of inspired oxygen applied, improves oxygenation and reduces mortality rate at 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Respiratory Distress Syndrome (ARDS) according to the American-European Consensus Conference definition, after 24 hours under mechanical ventilation.

Exclusion Criteria:

* Younger than 18-year-old
* Pregnancy
* Neuromuscular diseases
* Intracranial hypertension. Head trauma
* Left ventricular dysfunction
* Mechanical ventilation for more than 72 hours
* Previous barotrauma
* Patients with terminal stage of an illness and high risk of mortality within 90 days
* Patients who refused to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Arterial Oxygenation | 28 days
  Evolution of arterial oxygenation during the 28 days after study randomization

SECONDARY OUTCOMES:
Mortality | 28 days
  Mortality 28 days after randomization
Number of ventilator-free days at day 28 | 28 days
  Number of ventilator-free days at day 28 after randomization
multivariate analysis of mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: María del Consuelo Pintado, MD, PhD, Principal Investigator — Critical Care Unit. Universitary Hospital Principe de Asturias; Raúl de Pablo, MD, PhD, Principal Investigator — Critical Care Unit. Universitary Hospital Principe de Asturias
Locations (1):
- Critical Care Unit. Universitary Hospital Principe de Asturias, Alcalá de Henares, Madrid, Spain

REFERENCES:
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Suter PM, Fairley HB, Isenberg MD. Effect of tidal volume and positive end-expiratory pressure on compliance during mechanical ventilation. Chest. 1978 Feb;73(2):158-62. doi: 10.1378/chest.73.2.158. PMID 340159
- [Derived] Pintado MC, de Pablo R, Trascasa M, Milicua JM, Rogero S, Daguerre M, Cambronero JA, Arribas I, Sanchez-Garcia M. Individualized PEEP setting in subjects with ARDS: a randomized controlled pilot study. Respir Care. 2013 Sep;58(9):1416-23. doi: 10.4187/respcare.02068. Epub 2013 Jan 29. PMID 23362167